CLINICAL TRIAL: NCT01715649
Title: Evaluation of a Telehealth Intervention Combining Structured Self-Monitoring of Blood Glucose and Nurse Care Coordination Among People With Type 2 Diabetes Noninsulin-Treated
Brief Title: Telehealth Remote Patient Monitoring Study in People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sutter Health (Other)
Collaborators: LifeScan (Industry); GE Healthcare (Industry); University of California, Davis (Other)
Responsible Party: Principal Investigator, Deborah Greenwood, Diabetes Clinical Nurse Specialist, Sutter Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1208042ex
Record Dates: First submitted 2012-10-20; First posted 2012-10-29 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; self-management; remote patient monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Patient Education as Topic; Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control-usual care (No Intervention): Nurse care coordination in a telephonic diabetes disease management program
- Intervention paired testing and remote monitoring (Experimental): Telehealth remote patient monitoring, structured blood glucose and usual care Paired testing-weekly remote monitoring Data analysis Virtual visits in EHR
  Interventions: Behavioral: Patient education, self-monitoring of blood glucose and remote patient monitoring of blood glucose

INTERVENTIONS:
Behavioral: Patient education, self-monitoring of blood glucose and remote patient monitoring of blood glucose — In the intervention arm you will test your blood glucose 2 times a day (before and after a meal, activity or other event) using the glucose meter provided to you for use in this study and connect it to the Telehealth Unit. Every week the study team will review your blood glucose levels through the remote patient monitoring secure portal and send you a reminder through the Telehealth Unit with suggestions based on your blood glucose patterns. Once every month a study nurse will call you to review your blood glucose goals and discuss how you may be able to make changes in your health behaviors to improve your blood glucose levels. The study team will work with you to help you make changes to your behaviors that may improve your blood glucose.
  Arms: Intervention paired testing and remote monitoring

SUMMARY:
Telehealth remote patient monitoring is a means of using communications technology - such as telephones, computers, and the Internet - to connect patients remotely with their healthcare team from their homes. The investigators hope to learn more about improving healthy behaviors and blood glucose among persons with diabetes using telehealth remote patient monitoring technology to connect directly with nurse care coordinators.

The purpose of this study is to evaluate a process for improving blood glucose and healthy behaviors among people with type 2 diabetes using telehealth remote patient monitoring technology with nurse care coordinators. Some of the people in this study will work with a nurse care coordinator who will review your blood glucose weekly and call you at home every month for 3 months, while some of the people in this study will simply receive their normal care. At the end of the study, every participant will be asked questions about how they feel about their health care.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in diabetes disease management program
* ages 30-70
* HbA1c between 7.5% and 10.9% in the previous six months
* an Internet or 3G connection and email address;
* a working phone line (land line or cellular); and
* ability to read and understand the English language.

Exclusion Criteria:

* taking insulin;
* inability to independently engage in self-management behaviors (diagnosis of dementia, severe depression, schizophrenia, or cognitive impairment);
* severe complications, which would preclude achieving an HbA1c goal of 7% including diagnosis of the following:
* severe stroke;
* heart failure;
* end-stage renal disease;
* kidney dialysis; and
* legally blind.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Change from baseline to 6 months
  Lab test

SECONDARY OUTCOMES:
Empowerment | Change from baseline to 3 months
  Diabetes Empowerment Scale completed by survey
Behavior Change | Change from baseline to 3 months
  Summary of Diabetes Self-Care Behaviors scale completed by survey
Knowledge | Change from baseline to 3 months
  Michigan Diabetes Knowledge Test completed by survey

OTHER OUTCOMES:
Feasibility of incorporating the intervention into the existing program | 3 months
  Will include # of participants that complete intervention, #of nurse hours required to analyze data and interact with participant,and number of technology issues impacting use
Participant engagement with telehealth technology | 3 months
  # of participants that complete the 12 week program, # of participants that upload the blood glucose meter values to the technology

CONTACTS AND LOCATIONS:
Locations (1):
- Sutter Health, Sacramento, California, United States

REFERENCES:
- [Derived] Greenwood DA, Blozis SA, Young HM, Nesbitt TS, Quinn CC. Overcoming Clinical Inertia: A Randomized Clinical Trial of a Telehealth Remote Monitoring Intervention Using Paired Glucose Testing in Adults With Type 2 Diabetes. J Med Internet Res. 2015 Jul 21;17(7):e178. doi: 10.2196/jmir.4112. PMID 26199142